CLINICAL TRIAL: NCT07325981
Title: Effect of Biofeedback-Enhanced Exergaming, Exergaming Alone, and Traditional Physical Therapy on Motor Function, Adherence, and Engagement in Children With Cerebral Palsy (GMFCS I-II): A Randomized Controlled Trial
Brief Title: Effect of Biofeedback-Enhanced Exergaming, Exergaming Alone, and Traditional Physical Therapy on Motor Function, Adherence, and Engagement in Children With Cerebral Palsy: A RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Sajid Iqbal, Assistant Professor/Physical Therapist, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11120925SIPT
Record Dates: First submitted 2025-12-11; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy, exergaming, bio-feedback, GMFCS, traditional physical therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: In this experimental study design, participants will be randomly assigned to one of three separate intervention groups: exergaming, biofeedback-enhanced exergaming, and traditional physical therapy. Each group will receive only one intervention throughout the entire study period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exergaming (Experimental): The exergaming program will use Kinect Adventures (River Rush, Reflex Ridge) to train balance, agility, and trunk control; Kinect Sports to improve lower-limb activation, hand-eye coordination, and bilateral movements; Just Dance Kids for rhythmic stepping; and Kinect Party/Happy Action Theater to encourage free movement. Optional MIRA Rehab modules may target posture and agility. Sessions will be held three times per week for twelve weeks, starting with a light warm-up, followed by 20-30 minutes of targeted exergames, and ending with a cool-down. Game difficulty will progressively increase, and therapists will track progress through scores and completion times.
  Interventions: Other: exergaming
- biofeedback-enhanced exergaming (Experimental): This group will perform the same exergaming activities as the exergaming group, with the added integration of real-time multimodal biofeedback to enhance motor learning. The frequency and duration of sessions will be identical to the exergaming group. Participants will receive on-screen visual guides that indicate whether their movements are being performed correctly, along with auditory feedback through performance-linked cues such as pitch changes or sound alerts prompting postural adjustments. Optional vibration alerts from wearable devices may also be used to correct improper posture. The biofeedback system will incorporate surface EMG (Delsys Trigno) to assess bilateral muscle activity during gameplay, and motion tracking through the Microsoft Kinect SDK (v2 or Azure) to capture and analyze joint movements, posture, and detailed ranges of motion.
  Interventions: Other: biofeedback-enhanced exergaming
- traditional physical therapy (Active Comparator): Children in this group will receive standard physical therapy to improve gross motor function, especially balance and mobility. Sessions will be held three times per week for twelve weeks, lasting 30-45 minutes. The protocol includes a 5-minute warm-up, 12-15 minutes of strengthening for hip, knee, and ankle muscles, 8-10 minutes of balance training using wobble boards or foam, and 8-10 minutes of functional mobility tasks such as sit-to-stand and stair practice, followed by a 2-5 minute cool-down. Therapists will follow standardized instructions, and treatment fidelity will be monitored through checklists, with 10% of sessions audited monthly.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: exergaming — The exergaming program will use Kinect Adventures (River Rush, Reflex Ridge) for balance and agility, Kinect Sports for lower-limb activation and coordination, Just Dance Kids for rhythmic stepping, and Kinect Party/Happy Action Theater for free movement. Optional MIRA Rehab modules may target posture and agility. Sessions will occur three times weekly for twelve weeks, beginning with a light warm-up, followed by 20-30 minutes of targeted exergames, and ending with a cool-down. Game difficulty will increase as children improve, and therapists will track progress using scores and completion times.
  Arms: exergaming
Other: biofeedback-enhanced exergaming — This group will perform the same exergames as Intervention 1 but with real-time visual, auditory, and optional vibration feedback to enhance motor learning. Surface EMG (Delsys Trigno) will record bilateral muscle activity, and Microsoft Kinect SDK (v2/Azure) will track joint motion and posture. Session frequency and duration will be identical.
  Arms: biofeedback-enhanced exergaming
Other: Traditional Physical Therapy — Children in this group will receive standard physical therapy to improve gross motor function, especially balance and mobility. Sessions will be held three times per week for twelve weeks, lasting 30-45 minutes. The protocol includes a 5-minute warm-up, 12-15 minutes of strengthening for hip, knee, and ankle muscles, 8-10 minutes of balance training using wobble boards or foam, and 8-10 minutes of functional mobility tasks such as sit-to-stand and stair practice, followed by a 2-5 minute cool-down. Therapists will follow standardized instructions, and treatment fidelity will be monitored through checklists, with 10% of sessions audited monthly.
  Arms: traditional physical therapy

SUMMARY:
Cerebral Palsy (CP) accounts for approximately 0.9% of the global disease burden and affects 2.4-4% of children under 5 years old, with associated developmental and coordination impairments. Pediatric physical therapy aims to enhance independence and quality of life; however, maintaining adherence to conventional treatment remains a major challenge due to its repetitive and monotonous nature, leading to reduced motivation and limited functional progress.

Exergaming, integrating physical activity with interactive video games, has emerged as an engaging alternative shown to improve motor function, balance, and coordination in children with motor impairments. While existing evidence supports its effectiveness, few randomized studies have explored the addition of real-time physiological biofeedback (e.g., surface EMG with motion tracking) within exergaming platforms. Evidence on adherence and engagement outcomes also remains limited.

This trial addresses that gap by investigating the combined effects of biofeedback-enhanced exergaming versus exergaming alone and traditional physiotherapy in children with CP (GMFCS levels I-II). Incorporating real-time biofeedback provides immediate physiological feedback, potentially enhancing motor learning, motivation, and adherence, key components for improving long-term rehabilitation outcomes in pediatric populations.

DETAILED DESCRIPTION:
This single-blinded randomized controlled trial will be conducted at Ziauddin Hospital and the IHRI Rehabilitation Centre and School, Karachi, Pakistan. A total of 90 children (aged 6-12 years) with spastic diplegic or hemiplegic cerebral palsy (GMFCS levels I-II) will be recruited through purposive sampling and stratified by age band (6-8 vs. 9-12 years) and GMFCS level. Participants will be randomized (1:1:1) into three intervention groups using computer-generated permuted blocks with allocation concealment via sealed envelopes.

Outcome assessors and data analysts will be blinded. Inclusion requires adequate cognition (NIH Toolbox PSMT ≥ 25th percentile), functional mobility, and hearing/vision sufficient for exergaming tasks. Exclusion criteria include severe motor, cognitive, or sensory impairments, uncontrolled epilepsy, behavioral challenges, or concurrent clinical trial participation. The sample size (n=90) was determined via G*Power (effect size f=0.30, α=0.05, power=0.80) to detect clinically meaningful between-group differences in motor function (BOT-2).

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with Cerebral Palsy (CP), specifically spastic diplegia, spastic hemiplegia, or mild ataxia.

* Gross Motor Function Classification System (GMFCS) Level I or II.
* Male and female aged between 6 and 12 years at the time of enrollment.
* Manual Ability Classification System (MACS) Level I or II.
* Able to follow simple two-step commands, with or without augmentative and alternative communication (AAC).
* Demonstrates adequate cognitive functioning based on the NIH Toolbox Picture Sequence Memory Test (PSMT), scoring at or above the 25th percentile (T-score ≥ 40) based on age-adjusted norms.
* Hearing and vision adequate to participate in exergaming tasks (with or without assistive devices).
* Able to stand and participate in basic movements with or without minimal assistance.
* Willingness to participate and written informed consent from parent/guardian with assent from the child.

Exclusion Criteria:

* GMFCS Level III or higher, indicating significant gross motor limitations.

  * MACS Level III or higher, indicating significant manual impairment.
  * Severe uncorrected visual or hearing impairment that would interfere with interaction during exergaming.
  * Uncontrolled epilepsy or other neurological condition contraindicating active movement.
  * Significant behavioral or attention challenges that prevent engagement with game-based tasks.
  * Score below the 25th percentile on the PSMT, indicating insufficient episodic memory to follow game tasks.
  * Involvement in any other intervention trial that may interfere with study participation.
  * Medical conditions that contraindicate participation in physical activity (as determined by a physician).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Improvement | 4-6 months
  Outcome Measure Title:
  Gross Motor Function Measure (GMFM-88) total score (%)
  Description:
  Gross motor function will be assessed using the Gross Motor Function Measure-88 (GMFM-88), a standardized observational tool evaluating motor skills across five domains: lying & rolling, sitting, crawling & kneeling, standing, and walking/running/jumping. Scores are expressed as a percentage of the maximum possible score.
  Score range: 0-100% Interpretation: Higher scores indicate better gross motor function.
Balance Performance | 4-6 months
  Outcome Measure Title:
  Pediatric Balance Scale (PBS) total score
  Description:
  Balance performance will be measured using the Pediatric Balance Scale (PBS), a functional balance assessment adapted from the Berg Balance Scale. The scale consists of 14 tasks assessing static and dynamic balance during functional activities.
  Score range: 0-56 Interpretation: Higher scores indicate better balance performance.
Postural Control | 4-6 months
  Outcome Measure Title:
  Postural stability parameters derived from Kinect-based motion analysis
  Description:
  Postural control stability will be quantified using Kinect-based motion tracking, capturing center of mass displacement, joint angles, and sway during task-based activities. Movement stability indices (e.g., reduced sway amplitude and improved alignment) will be derived from kinematic data.
  Measurement units: Degrees (joint angles), millimeters (displacement), task-specific stability indices Interpretation: Lower sway and improved alignment indicate better postural stability.
Functional Mobility | 4-6 months
  Outcome Measure Title:
  Timed Up and Go (TUG) test duration (seconds)
  Description:
  Functional mobility will be assessed using the Timed Up and Go (TUG) test, which measures the time required to stand from a seated position, walk 3 meters, turn, return, and sit down.
  Score range: Continuous variable (seconds) Interpretation: Shorter completion times indicate better functional mobility.

SECONDARY OUTCOMES:
Muscle Activation Patterns | 4-6 months
  Outcome Measure Title:
  Surface electromyography (sEMG) amplitude and activation timing during task performance
  Description:
  Surface EMG will be used to record muscle activation amplitude and timing during functional tasks. Outcome variables will include normalized EMG amplitude and coordination patterns across target muscle groups.
  Measurement units: Microvolts (µV), normalized activation ratios Interpretation: More efficient and coordinated activation patterns indicate improved motor control.
Game performance score | 4-6 months
  Score range: System-generated scores Interpretation: Higher game scores indicate improved motor learning and performance.
task completion time during virtual-based tasks | 4-6 months
  Description:
  Motor learning including task completion time generated by the virtual rehabilitation system.
  Interpretation: reduced completion times indicate improved motor learning and performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Participant confidentiality and institutional policy restrict the sharing of individual-level data.